06/03/2025 v1.1

IRAS ID: 341922



IRAS ID: 341922

## **FACILITATOR CONSENT FORM**

Title of Project: A study to explore the feasibility and efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms

following a traumatic birthing experience. Name of Researcher: Grace Rodgers Please initial box I confirm that I have read the facilitator information sheet (version 1.1, dated 06/03/2025 for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I understand that my participation is voluntary and that I am free to withdraw at any time 2. without giving any reason. I understand that should I withdraw before the study has finished; any data already collected may be used in data analysis. 3. I understand that the information collected from me will be used to support other research in the future and may be shared anonymously with other researchers. I understand that my anonymised data will be used for dissemination in publications (e.g., within 4. scientific journals/conference abstracts). This might include anonymised quotes. 5. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature seeking consent (OPTIONAL) If you would like to receive the results of the study when it is complete, please provide your email address below: